CLINICAL TRIAL: NCT01754766
Title: AGN-229666 for the Treatment of Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 229666-002
Record Dates: First submitted 2012-12-19; First posted 2012-12-21 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2013-12

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- AGN-229666 Dose A (Experimental): One drop of AGN-229666 Dose A into each eye on Day 1 and Day 15.
  Interventions: Drug: AGN-229666
- AGN-229666 Dose B (Experimental): One drop of AGN-229666 Dose B into each eye on Day 1 and Day 15.
  Interventions: Drug: AGN-229666
- vehicle of AGN-229666 (Placebo Comparator): One drop of vehicle of AGN-229666 into each eye on Day 1 and Day 15.
  Interventions: Other: vehicle of AGN-229666

INTERVENTIONS:
Drug: AGN-229666 — One drop of AGN-229666 into each eye on Day 1 and Day 15.
  Arms: AGN-229666 Dose A; AGN-229666 Dose B
Other: vehicle of AGN-229666 — One drop of vehicle of AGN-229666 into each eye on Day 1 and Day 15.
  Arms: vehicle of AGN-229666

SUMMARY:
This study will evaluate the safety and efficacy of AGN-229666 for the treatment of allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients living in Japan with a history of allergic conjunctivitis
* Willing to discontinue wearing contact lenses during the study period

Exclusion Criteria:

* Use of nicotine products during the study period
* Presence of active eye infection (bacterial, viral, or fungal)
* History of an ocular herpetic infection
* Eye surgery intervention within 3 months and/or a history of refractive surgery within the past 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AGN-229666 Dose A | AGN-229666 Dose B | Vehicle of AGN-229666
Started | 31 | 29 | 30
Completed | 30 | 28 | 30
Not Completed | 1 | 1 | 0
Not completed — Personal reasons | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-229666 Dose A | AGN-229666 Dose B | Vehicle of AGN-229666 | Total
Number analyzed (Participants) | 31 | 29 | 30 | 90
Age, Customized [Number; unit: Participants]
  20-30 years | 11 | 7 | 4 | 22
  >30-40 years | 7 | 7 | 10 | 24
  >40 years | 13 | 15 | 16 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 15 | 44
  Male | 17 | 14 | 15 | 46

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching Score at Day 1
Description: The participant evaluated ocular itching in both eyes 5 minutes post conjunctival allergen challenge (CAC) (8 hours post-dose) at Day 1 using a 9-point scale in half-unit increments where: 0=none to 4=incapacitating itch with an irresistible urge to rub. The score for each participant was the average of the score of both eyes.
Time Frame: Day 1
Population: Modified Intent-to-treat (MITT) population included all randomized participants with ocular itching score data available for this time point
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AGN-229666 Dose A | AGN-229666 Dose B | Vehicle of AGN-229666
Number analyzed (Participants) | 31 | 29 | 30
Score on a scale | 0.500 (0.5123) | 0.319 (0.3947) | 1.867 (0.9485)

2. Secondary Outcome: Ocular Itching Score at Day 15
Description: The participant evaluated ocular itching in both eyes 5 minutes post conjunctival allergen challenge (16 hours post-dose) at Day 15 using a 9-point scale in half-unit increments where: 0=none to 4=incapacitating itch with an irresistible urge to rub. The score for each participant was the average of the score of both eyes.
Time Frame: Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AGN-229666 Dose A | AGN-229666 Dose B | Vehicle of AGN-229666
Number analyzed (Participants) | 30 | 28 | 30
Score on a scale | 0.358 (0.4083) | 0.214 (0.3582) | 1.258 (0.9249)

3. Secondary Outcome: Conjunctival Hyperemia Score
Description: Conjunctival hyperemia is the engorgement of the blood vessels (redness) of the clear membrane covering the white surface of the eye. Conjunctival hyperemia was evaluated 15 minutes post conjunctival allergen challenge (CAC) (8 hours post dose) on Day 1 for both eyes using a 9-point scale in half-unit increments where: 0=none to 4=Extremely severe. The score for each participant was the average of the score of both eyes.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AGN-229666 Dose A | AGN-229666 Dose B | Vehicle of AGN-229666
Number analyzed (Participants) | 31 | 29 | 30
Score on a scale | 1.387 (0.6118) | 1.345 (1.0531) | 1.633 (0.5972)

ADVERSE EVENTS:
Arm/Group | AGN-229666 Dose A | AGN-229666 Dose B | Vehicle of AGN-229666
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 2/29 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-229666 Dose A (N=31) | AGN-229666 Dose B (N=29) | Vehicle of AGN-229666 (N=30)
Ocular hyperaemia (Eye disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.